CLINICAL TRIAL: NCT01684995
Title: Motivation and Nicotine Patch Treatment for Under-served Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: Quit_RIte_RI; R01DA010860 (NIH)
Record Dates: First submitted 2012-08-29; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal (Active Comparator): Brief physician advice to quit smoking plus nicotine patch
  Interventions: Behavioral: Brief physician advice; Drug: nicotine patch
- Tailored (Experimental)
  Interventions: Behavioral: Brief physician advice; Drug: nicotine patch; Behavioral: Individually Tailored Behavioral Skills training

INTERVENTIONS:
Behavioral: Brief physician advice — Brief physician advice to quit smoking
Drug: nicotine patch — nicotine patch
Behavioral: Individually Tailored Behavioral Skills training — Individually tailored behavioral skills training for smoking cessation
  Arms: Tailored

SUMMARY:
The goal of this study is to test, in combination with the nicotine patch, the incremental efficacy of a motivationally tailored behavioral intervention over a minimal intervention. The interventions will be delivered through primary care medical clinics. The defined population comprises low income, less educated smokers who will vary in their level of motivation to quit smoking. Patients will be randomly assigned within clinics to one of two interventions (a) Nicotine patch prescription plus brief physician advice (minimal care); and (b) Nicotine patch prescription plus brief physician advice, with the addition of a tailored motivational intervention, a behavioral skills counseling session for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently smoking at least 10 cigarettes/day for past 3 months
* Speak English or Spanish
* Have a telephone or live close to a relative or neighbor with a telephone
* Agree to participate in the study and be available over the next 6 months.

Exclusion Criteria:

* Unable to use nicotine patch due to medical status
* Active skin condition or history of skin allergy
* Currently using smokeless tobacco, nicotine replacement or other smoking cessation treatment
* Pregnant or nursing

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1996-12; Primary Completion 1999-11 (Actual); Study Completion 1999-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Bock B, Lopes CE, van den Berg JJ, Roberts MB, Stein LA, Martin RA, Martin SA, Clarke JG. Social support and smoking abstinence among incarcerated adults in the United States: a longitudinal study. BMC Public Health. 2013 Sep 17;13:859. doi: 10.1186/1471-2458-13-859. PMID 24044880